CLINICAL TRIAL: NCT02936401
Title: Interventions for Symptom Management in Older Patients With HAND
Brief Title: Mindfulness Based Stress Reduction for Older Adults With HIV Associated Neurocognitive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Harvard School of Public Health (HSPH) (Other); Northwestern University (Other); University of Missouri, St. Louis (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01NR015223 (NIH); R01NR015223 (NIH)
Record Dates: First submitted 2016-07-27; First posted 2016-10-18 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Impaired Cognition; HIV Infection
MeSH Terms: conditions — Cognition Disorders; HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR (Experimental): Participants in this arm enter the 8-week MBSR course immediately after the baseline visit.
  Interventions: Behavioral: MBSR
- CONTROL (Experimental): Participants in the waitlist control arm will receive standard of care for 16 weeks after the baseline visit, and then will be offered an identical 8-week MBSR course.
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Mindfulness Based Stress Reduction (MBSR) is a standardized 8 week course taught by trained instructors.

SUMMARY:
The purpose of this study is to determine the efficacy of Mindfulness Based Stress Reduction (MBSR) to alleviate stress, anxiety, and depressive symptoms, and improve attention among patients aged 60 or older who suffer from HIV-associated neurocognitive disorders (HAND) and have maximized treatment options.

DETAILED DESCRIPTION:
This study addresses symptom management for patients aged 60 and older who are living with HIV infection, are on combination antiretroviral therapy (cART) with suppressed viral loads, and yet continue to experience behavioral and cognitive symptoms of HIV-associated neurocognitive disorders (HAND). It is increasingly relevant that HAND persists despite cART, impacting between 30-50% of elders living with HIV. Patients suffer symptoms that are pervasive in their impact on everyday functioning and quality of life; yet these patients are currently left with a dearth of treatment options. In this study, the investigators employ a randomized controlled evaluation of Mindfulness Based Stress Reduction (MBSR) to target attention, stress, anxiety, and depressive symptoms among patients who have HAND and have maximized treatment options. The investigators will employ intrinsic connectivity network (ICN) analyses of resting state functional magnetic resonance imaging to demonstrate increased strength of brain networks corresponding to improved symptoms. The investigators will quantify social networks and perceived strength of social networks to determine if they moderate the main findings. Together this work employs geriatric, neuroscience and complementary medicine disciplines to reduce the symptom burden in aging HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* HIV-infected. For cases in which a participant has an undetectable plasma viral load and is not currently on cART, the participant will be asked to complete HIV antibody testing.
* Undetectable plasma viral load
* Symptomatic and sufficient neuropsychological testing abnormality to be rated as having impairment by consensus conference, but deficits in everyday functioning that would rate them as having no more than moderate disease. Participants with severe deficits consistent with dementia will not be randomized unless the study team agrees that deficits are mild enough to withstand rigors of MBSR.

Exclusion Criteria:

* Age < 55 years
* Failure to attend screening visits after two attempts and despite support offered
* Unwilling to participate in 8-week intervention
* Endorsing illicit drug use in the past 6 months
* Current or extensive previous mindfulness practitioner
* Detectable plasma HIV RNA (VL) in the previous 6 months or at enrollment. Individuals with VL <500 copies will be allowed to enroll if they have a history of UD VL with unchanged cART and show documentation of their past two clinical VL at UD levels (so called "viral blips").
* Any treatable condition that may impact cognition, including:

  * Neurosyphilis (cases with serum RPR positive will undergo lumbar puncture to evaluate)
  * Thyroid disorders (untreated)
  * B12 deficiency (untreated)
  * Cancer (requiring chemotherapy)
  * Neurological or psychiatric conditions where treatment options exist, such as multiple sclerosis, schizophrenia, uncontrolled epilepsy, recent and untreated major depression
  * HIV CNS escape (lumbar punctures will be completed in cases with clinical scenarios worrisome for escape as done clinically; e.g. more rapid course, new neurological symptoms, recent resistance in plasma)
* Language other than English as the main language of oral and written communication
* Inability to provide informed consent or assent with a legal surrogate to sign consent
* Major recent head injury, stroke, or major confounding cognitive factors including:

  * Cognitive impairment caused primarily by alcohol or substance use
  * Current active use of methamphetamine, cocaine or illicit use of narcotics (determined at screening and enrollment visits via clinical interview of substance abuse and dependence criteria)
  * MRI demonstrating current or past CNS lesions deemed to be clinically significant including that from past opportunistic infections but excluding white matter injury, as can be seen with cerebrovascular disease
  * Active brain infection, except for HIV
  * Significant systemic medical illness such as cancer requiring chemotherapy or end-stage cardiac or renal insufficiency
* Unstable psychiatric condition (e.g. active psychosis, suicidal ideation, homicidal ideation) or mental health or medical condition that, in the opinion of the investigators, will make it difficult for the potential participant to participate in the intervention
* Cases where the investigators feel the participant won't be able to complete the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Continuous Performance Task | 48 weeks after enrollment
  A neuropsychological test to assess attention and information processing and executive functioning
Symbol-Digit modalities test | 48 weeks after enrollment
  A neuropsychological test to assess executive functioning
Letter Number Sequencing | 48 weeks after enrollment
  A neuropsychological test to assess executive functioning
Activities of Daily Living (ADL) & Instrumental Activities of Daily Living (IADL) scales | 48 weeks after enrollment
  Questionnaires to assess everyday function
Perceived Stress Scale | 48 weeks after enrollment
  Questionnaire to assess stress
State-Trait Anxiety Inventory | 48 weeks after enrollment
  Questionnaire to assess anxiety
Geriatric Depression Scale | 48 weeks after enrollment
  Questionnaire to assess depression
Buss-Durkee Irritability subscale | 48 weeks after enrollment
  Questionnaire to assess irritability
Center for Neurological Study - Lability Scale | 48 weeks after enrollment
  Questionnaire to assess affective lability
Affective Intensity Measure | 48 weeks after enrollment
  Questionnaire to assess euphoria
World Health Organization Quality of Life - HIV Scale | 48 weeks after enrollment
  Questionnaire to assess quality of life
Connectivity of the default mode network (DMN) as determined by analysis of resting state functional magnetic resonance imaging | 16 weeks after enrollment
Connectivity of the salience network (SAL) as determined by analysis of resting state functional magnetic resonance imaging | 16 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Victor Valcour, MD PhD, Principal Investigator — University of California, San Francisco; Judith Moskowitz, PhD MPH, Principal Investigator — Northwestern University
Locations (1):
- UCSF Memory and Aging Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson KR, Smurzynski M, Parsons TD, Wu K, Bosch RJ, Wu J, McArthur JC, Collier AC, Evans SR, Ellis RJ. The prevalence and incidence of neurocognitive impairment in the HAART era. AIDS. 2007 Sep 12;21(14):1915-21. doi: 10.1097/QAD.0b013e32828e4e27. PMID 17721099
- [Background] Kanmogne GD, Kuate CT, Cysique LA, Fonsah JY, Eta S, Doh R, Njamnshi DM, Nchindap E, Franklin DR Jr, Ellis RJ, McCutchan JA, Binam F, Mbanya D, Heaton RK, Njamnshi AK. HIV-associated neurocognitive disorders in sub-Saharan Africa: a pilot study in Cameroon. BMC Neurol. 2010 Jul 13;10:60. doi: 10.1186/1471-2377-10-60. PMID 20626870
- [Background] Valcour V, Shikuma C, Shiramizu B, Watters M, Poff P, Selnes O, Holck P, Grove J, Sacktor N. Higher frequency of dementia in older HIV-1 individuals: the Hawaii Aging with HIV-1 Cohort. Neurology. 2004 Sep 14;63(5):822-7. doi: 10.1212/01.wnl.0000134665.58343.8d. PMID 15365130
- [Background] Tozzi V, Balestra P, Bellagamba R, Corpolongo A, Salvatori MF, Visco-Comandini U, Vlassi C, Giulianelli M, Galgani S, Antinori A, Narciso P. Persistence of neuropsychologic deficits despite long-term highly active antiretroviral therapy in patients with HIV-related neurocognitive impairment: prevalence and risk factors. J Acquir Immune Defic Syndr. 2007 Jun 1;45(2):174-82. doi: 10.1097/QAI.0b013e318042e1ee. PMID 17356465
- [Background] Sacktor N, McDermott MP, Marder K, Schifitto G, Selnes OA, McArthur JC, Stern Y, Albert S, Palumbo D, Kieburtz K, De Marcaida JA, Cohen B, Epstein L. HIV-associated cognitive impairment before and after the advent of combination therapy. J Neurovirol. 2002 Apr;8(2):136-42. doi: 10.1080/13550280290049615. PMID 11935465
- [Background] Cysique LA, Brew BJ. Neuropsychological functioning and antiretroviral treatment in HIV/AIDS: a review. Neuropsychol Rev. 2009 Jun;19(2):169-85. doi: 10.1007/s11065-009-9092-3. Epub 2009 May 9. PMID 19424802
- [Background] Cysique LA, Maruff P, Brew BJ. Variable benefit in neuropsychological function in HIV-infected HAART-treated patients. Neurology. 2006 May 9;66(9):1447-50. doi: 10.1212/01.wnl.0000210477.63851.d3. PMID 16682686
- [Background] Vance DE, Fazeli PL, Grant JS, Slater LZ, Raper JL. The role of neuroplasticity and cognitive reserve in aging with HIV: recommendations for cognitive protection and rehabilitation. J Neurosci Nurs. 2013 Oct;45(5):306-16. doi: 10.1097/JNN.0b013e31829d8b29. PMID 24025470
- [Background] Cohen-Katz J, Wiley S, Capuano T, Baker DM, Deitrick L, Shapiro S. The effects of mindfulness-based stress reduction on nurse stress and burnout: a qualitative and quantitative study, part III. Holist Nurs Pract. 2005 Mar-Apr;19(2):78-86. doi: 10.1097/00004650-200503000-00009. PMID 15871591
- [Background] Moynihan JA, Chapman BP, Klorman R, Krasner MS, Duberstein PR, Brown KW, Talbot NL. Mindfulness-based stress reduction for older adults: effects on executive function, frontal alpha asymmetry and immune function. Neuropsychobiology. 2013;68(1):34-43. doi: 10.1159/000350949. Epub 2013 Jun 15. PMID 23774986
- [Background] Gayner B, Esplen MJ, DeRoche P, Wong J, Bishop S, Kavanagh L, Butler K. A randomized controlled trial of mindfulness-based stress reduction to manage affective symptoms and improve quality of life in gay men living with HIV. J Behav Med. 2012 Jun;35(3):272-85. doi: 10.1007/s10865-011-9350-8. Epub 2011 May 20. PMID 21597980
- [Background] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Background] Carmody J, Baer RA. Relationships between mindfulness practice and levels of mindfulness, medical and psychological symptoms and well-being in a mindfulness-based stress reduction program. J Behav Med. 2008 Feb;31(1):23-33. doi: 10.1007/s10865-007-9130-7. Epub 2007 Sep 25. PMID 17899351
- [Background] Jain S, Shapiro SL, Swanick S, Roesch SC, Mills PJ, Bell I, Schwartz GE. A randomized controlled trial of mindfulness meditation versus relaxation training: effects on distress, positive states of mind, rumination, and distraction. Ann Behav Med. 2007 Feb;33(1):11-21. doi: 10.1207/s15324796abm3301_2. PMID 17291166
- [Background] Shapiro SL, Oman D, Thoresen CE, Plante TG, Flinders T. Cultivating mindfulness: effects on well-being. J Clin Psychol. 2008 Jul;64(7):840-62. doi: 10.1002/jclp.20491. PMID 18484600
- [Background] Cohen-Katz J, Wiley SD, Capuano T, Baker DM, Kimmel S, Shapiro S. The effects of mindfulness-based stress reduction on nurse stress and burnout, Part II: A quantitative and qualitative study. Holist Nurs Pract. 2005 Jan-Feb;19(1):26-35. doi: 10.1097/00004650-200501000-00008. PMID 15736727